CLINICAL TRIAL: NCT01681446
Title: The Effect of Postoperative Interferon-alpha Treatment in Patients Underwent Curative Surgery for Hepatocellular Carcinoma With a Low miR-26 Expression: a Multi-center Randomized Clinical Trial.
Brief Title: Adjuvant IFN-α for Patients Underwent Curative Surgery for HCC With a Low miR-26 Expression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jia Fan, Professor of Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCI IFNa miR-26
Record Dates: First submitted 2012-08-23; First posted 2012-09-10 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; interferon-alpha; miR-26
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Interferon-alpha; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interferon-alpha (IFN-alpha) (Active Comparator): interferon-alpha is intramuscularly or subcutaneously injected at 30 μg three times a week or 50 μg twice a week for 18 months
  Interventions: Drug: interferon-alpha (IFN-alpha)
- control (No Intervention): no anti-cancer interventions were assigned

INTERVENTIONS:
Drug: interferon-alpha (IFN-alpha) — interferon-alpha is intramuscular injected 30 μg three times a week or 50 μg twice a week for 18 months
  Other Names: Recombinant Human Interferon α1b for Injection; SINOGEN
  Arms: interferon-alpha (IFN-alpha)

SUMMARY:
The purpose of the study is to determine whether interferon-alpha is effective in prevention of tumor recurrence for the patients with a low miR-26 expression in tumor after curative resection of hepatocellular carcinoma.

DETAILED DESCRIPTION:
BACKGROUND: Postoperative interferon-alpha (IFN-alpha) therapy improved survival in patients with hepatocellular carcinoma (HCC). MiR-26 is a predictive marker for the effect of postoperative interferon-alpha treatment in patients with HCC. Our study is to identify the effect of postoperative IFN-alpha treatment in patients with a low miR-26 expression in tumor after resection of HCC.

METHODS: A quantitative RT-PCR assays of miR-26 are performed on specimens which are collected from patients who underwent a curative resection of HCC. These patients with low miR-26 expression will return to the hospital 4 to 6 weeks after the resection following the baseline examination to rule out residual tumor. If all requirements are satisfied, these patients will be randomly assigned to the treatment group who received postoperative IFN-alpha therapy or the control group who will not receive any anti-cancer treatment. Disease-free survival, overall survival, time to recurrence and the side effects will be observed.

Anticipated RESULTS: IFN-alpha treatment improved the disease-free survival in patients with a low miR-26 expression in tumor after curative resection of HCC, probably by inhibiting tumor recurrence.

ELIGIBILITY:
Perioperative Period Inclusion Criteria:

1. Signed informed consent;
2. Aged ≥ 18 years and ≤ 75 years old, male or female；
3. Patients with a low miR-26 expression in tumor (confirmed by RT-PCR) underwent a curative resection of HCC;
4. The tumor characteristics must meet the following:

   1. tumor diameter is between 3 to 8 centimeters,and the number of tumor is less than 3
   2. no thrombosis is detected in the main branches of the portal vein, hepatic vein and bile duct by preoperative imaging or by intra-operative findings
   3. no extrahepatic and lymph node metastasis

Perioperative Period Exclusion Criteria:

1. Concomitant malignant primary tumor(s) in other systems is/are present;
2. The subject receives any previous systemic anti-HCC therapy prior to the resection surgery, such as liver transplantation, intervention, ablation, radiotherapy, chemotherapy, molecular targeted therapy or other anti-HCC therapy;
3. The subject takes other study/investigational drugs during this study;
4. The subject has cerebrovascular accident, renal insufficiency, depression, hyperthyreosis, hypothyroidism or other severe uncontrolled diseases;
5. The subject has a history of study drug or similar drug allergy.

Baseline (Post-Surgery 4 to 6 weeks) Inclusion Criteria:

1. Baseline (post-resection) blood routine examination shows that the number of leukocyte>2.5*10^9/L and platelet count>40*10^9/L;
2. Child-Pugh score of class A at baseline.

Baseline (Post-Surgery 4 to 6 weeks) Exclusion Criteria:

1. Concomitant malignant primary tumor(s) in other systems is/are present;
2. The subject takes other study/investigational drugs within 4 weeks prior to randomization;
3. The baseline examination indicates that infection, bleeding, bile leakage, or other postoperative complications are present;
4. The baseline examination suggests the presence of tumor metastasis;
5. The subject has cerebrovascular accident, renal insufficiency, depression, hyperthyreosis, hypothyroidism or other severe uncontrolled diseases;
6. The subject has a history of investigational drug or similar drug allergy;
7. The subject is pregnant, lactating, or urine pregnancy test result is positive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2012-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years
  interval between the dates of surgery and tumor recurrence or patient death

SECONDARY OUTCOMES:
overall survival | 5 years
  interval between the dates of surgery and patient death
time to recurrence | 5 years
  interval between the dates of surgery and tumor recurrence
Number of Participants with Adverse Events | eighteen months
  Number of Participants with Adverse Events（hypohepatia,fever,leukopenia and thrombopenia）will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD, PHD, Principal Investigator — Liver Cancer Institute and Zhongshan Hospital, Fudan University, Shanghai, China; Xin Wei Wang, PhD, Principal Investigator — National Cancer Institute, NIH, US
Locations (5):
- China (5):
  - The Mengchao hepatobiliary hospital，Fujian Medical University，and Liver disease research center of Fujian province, Fuzhou, Fujian
  - Zhongshan Hospital, Xiamen University, Xiamen, Fujian
  - Liver Cancer Institute and Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - ShanghaiBio Coorperation, Shanghai, Shanghai Municipality
  - Tumor Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality

REFERENCES:
- [Background] Ji J, Shi J, Budhu A, Yu Z, Forgues M, Roessler S, Ambs S, Chen Y, Meltzer PS, Croce CM, Qin LX, Man K, Lo CM, Lee J, Ng IO, Fan J, Tang ZY, Sun HC, Wang XW. MicroRNA expression, survival, and response to interferon in liver cancer. N Engl J Med. 2009 Oct 8;361(15):1437-47. doi: 10.1056/NEJMoa0901282. PMID 19812400
- [Background] Sun HC, Tang ZY, Wang L, Qin LX, Ma ZC, Ye QH, Zhang BH, Qian YB, Wu ZQ, Fan J, Zhou XD, Zhou J, Qiu SJ, Shen YF. Postoperative interferon alpha treatment postponed recurrence and improved overall survival in patients after curative resection of HBV-related hepatocellular carcinoma: a randomized clinical trial. J Cancer Res Clin Oncol. 2006 Jul;132(7):458-65. doi: 10.1007/s00432-006-0091-y. Epub 2006 Mar 24. PMID 16557381
- [Background] Lo CM, Liu CL, Chan SC, Lam CM, Poon RT, Ng IO, Fan ST, Wong J. A randomized, controlled trial of postoperative adjuvant interferon therapy after resection of hepatocellular carcinoma. Ann Surg. 2007 Jun;245(6):831-42. doi: 10.1097/01.sla.0000245829.00977.45. PMID 17522506
- [Background] Clavien PA. Interferon: the magic bullet to prevent hepatocellular carcinoma recurrence after resection? Ann Surg. 2007 Jun;245(6):843-5. doi: 10.1097/SLA.0b013e31805d0788. No abstract available. PMID 17522507
- [Background] Qian YB, Zhang JB, Wu WZ, Fang HB, Jia WD, Zhuang PY, Zhang BH, Pan Q, Xu Y, Wang L, Tang ZY, Sun HC. P48 is a predictive marker for outcome of postoperative interferon-alpha treatment in patients with hepatitis B virus infection-related hepatocellular carcinoma. Cancer. 2006 Oct 1;107(7):1562-9. doi: 10.1002/cncr.22206. PMID 16948122
- [Background] Wang L, Tang ZY, Qin LX, Wu XF, Sun HC, Xue Q, Ye SL. High-dose and long-term therapy with interferon-alfa inhibits tumor growth and recurrence in nude mice bearing human hepatocellular carcinoma xenografts with high metastatic potential. Hepatology. 2000 Jul;32(1):43-8. doi: 10.1053/jhep.2000.8525. PMID 10869287
- [Background] Wang L, Wu WZ, Sun HC, Wu XF, Qin LX, Liu YK, Liu KD, Tang ZY. Mechanism of interferon alpha on inhibition of metastasis and angiogenesis of hepatocellular carcinoma after curative resection in nude mice. J Gastrointest Surg. 2003 Jul-Aug;7(5):587-94. doi: 10.1016/s1091-255x(03)00072-6. PMID 12850669